CLINICAL TRIAL: NCT01913431
Title: A Multicenter, Double-blind, Active-controlled, Randomized, Parallel Group Study to Demonstrate the Comparison and Evaluation of Baracle Tab.® and Baraclude Tab.® for HBeAG Chronic Hepatitis B
Brief Title: Baracle Tab. ® Versus Baraclude Tab.® for Patients With HBeAg Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ETV_HB_IV
Record Dates: First submitted 2013-07-28; First posted 2013-08-01 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: HBeAg-Positive Chronic Hepatitis B
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baracle Tab.® (Experimental): (It can be also placebo) dosage: 2 tablets daily for 48 weeks
  Interventions: Drug: Baracle Tab.®
- Baraclude Tab.® (Experimental): (It can be also placebo) dosage: 2 tablets daily for 48 weeks
  Interventions: Drug: Baraclude Tab.®

INTERVENTIONS:
Drug: Baracle Tab.®
  Arms: Baracle Tab.®
Drug: Baraclude Tab.®
  Arms: Baraclude Tab.®

SUMMARY:
This is a multicenter, double blind, active-controlled, randomized, parallel group study to demonstrate the anti-viral activity and safety of Baracle Tab. and Baraclude Tab. for patients with HBeAg Chronic Hepatitis B. The subject will receive two tablets daily for 48 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with HbeAg Chronic Hepatitis B for at least six months starting from the Screening visit
* Subjects with HBsAg-Positive diagnosed at the screening visit
* Subjects with HBeAg-Positive or HBeAg-negative diagnosed at the screening visit
* For those who were diagnosed HBeAg-Positive, HBV DNA level should be equal or more than 1x10^5 copies/ml
* For those who were diagnosed HBeAg-Negative, HBV DNA level should be equal or more than 1x10^5 copies/ml
* Subjects who were NOT administrated any anti-viral agents including interferon or pegylated interferon

Exclusion Criteria:

* Subjects with HCV, HDV or HIV
* Subjects with decompensated liver disease who have more than 2.5mg/dl of total bilirubin, longer than 3 seconds of prothrombin time, less than 30g/l of serum albumin
* With medical history of hemorrhage, hepatic encephalopathy, or dyshepatia due to ascites, jaundice, varicose vein
* Less than 50ml/min of creatinine clearance diagnosed at the screening visit
* More than 50 ng/ml of alpha-fetoprotein at the screening visit
* Involved in other studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2015-11-06 (Actual); Study Completion 2015-11-06 (Actual)

PRIMARY OUTCOMES:
the Difference between HBV DNA level(log10) and the base line of HBV DNA level(log10) | 52 weeks
  measured at 24th week of the administration

SECONDARY OUTCOMES:
the percentage of participants who have less than 300 copies/ml of HBV DNA (undetectable titre) | 52 weeks
  measured at 24th/48th week of the administration
the proportion of participants with normalization of serum alanine aminotransferase (less than 1.0 times the upper limit of normal) | 52 weeks
  measured at 24th/48th week of the administration
the percentage of participants who have lost HBeAg | 52 weeks
  HBeAg of the participants was found positive at their screening visit. Also, the measurement performs 24th/48th week of the administration.

CONTACTS AND LOCATIONS:
Overall Officials: Han Chu Lee, M.D., Principal Investigator — Asan Medical Center; Si Hyun Bae, M.D, Principal Investigator — The Catholic University of Korea; Ju Hyun Kim, M.D., Principal Investigator — Gachon University of Medicine and Science Gil Medical Center; Jae Seok Hwang, M.D., Principal Investigator — Keimyung University Dongsan Medical Center; So Young Kwon, M.D., Principal Investigator — Konkuk University Hospital; Won Young Tak, Principal Investigator — Kyunpook National University Hospital; Jong Eun Yeon, M.D., Principal Investigator — Korae University Guro Hospital; Sang Young Han, M.D., Principal Investigator — Dong-A University Hospital; Joon Hyouk Lee, M.D., Principal Investigator — Samsung Medical Center; Jung Hwan Yoon, M.D., Principal Investigator — Seoul National University Hospital; Sang Hoon Ahn, M.D., Principal Investigator — Severance Hospital; Neung Hwa Park, M.D., Principal Investigator — Ulsan University Hospital; Youn Jae Lee, M.D., Principal Investigator — Inje University; In Hee Kim, M.D., Principal Investigator — Chonbuk National University Hospital; Byung Seok Lee, M.D., Principal Investigator — Chungnam National University Hospital
Locations (1):
- Asan Medical Center, Seoul, South Korea